CLINICAL TRIAL: NCT04578678
Title: Can Subthalamic Stimulation Using Directional Electrodes Improve Postoperative Management in Parkinson's Disease: A Post-market Study - Steeropt
Brief Title: Can Subthalamic Stimulation Using Directional Electrodes Improve Postoperative Management in Parkinson's Disease
Acronym: Steeropt
Status: Active, not recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-00475
Record Dates: First submitted 2020-09-08; First posted 2020-10-08 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Parkinson's Disease; Deep Brain Stimulation
Keywords: Apathy; Dysarthria; Neuropsychiatric Symptoms; Steering; Non-motor Symptoms; Motor State
MeSH Terms: conditions — Parkinson Disease; Lethargy; Dysarthria | interventions — ast-1 proteins, C elegans

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Apathy Group: Patients diagnosed with apathy
  Interventions: Other: Steering
- Dysarthria Group: Patients diagnosed with dysarthria
  Interventions: Other: Steering
- No Apathy and Dysarthria Group: Patients diagnosed with neither apathy nor dysarthria
- Apathy and Dysarthria Group: Patients diagnosed with apathy as well as dysarthria
  Interventions: Other: Steering

INTERVENTIONS:
Other: Steering — Fine tuning of the STN-DBS settings
  Groups: Apathy Group; Apathy and Dysarthria Group; Dysarthria Group

SUMMARY:
The primary objective of the study is to determine if subthalamic nucleus (STN) deep brain stimulation (DBS) using the Vercise directional leads improves neuropsychiatric state and neuropsychiatric fluctuations 12 months after surgery in a large consecutive series of STN-DBS Parkinson's disease (PD) patients.

DETAILED DESCRIPTION:
This project of further use of health-related data with consent by the participants is a prospective, international project to evaluate the improvement of neuropsychiatric symptoms and the quality of life 12 months after surgery in a large consecutive series of STN-DBS PD patients using novel implantable Neurostimulator Systems (Boston Scientific). The project will investigate if a fine tuning of the STN-DBS settings could alleviate neuropsychiatric fluctuations, apathy as well as DBS-induced dysarthria and global motor state. The tuning is performed in agreement with the instruction for use of all devices used. Further objectives are validation of new tools that are presently entering clinical routine in optimizing postoperative management like individual current sources, steering, imaging of volume of tissue activated, and beta-oscillations.

The data originates from patients suffering from levodopa-responsive PD which are not adequately controlled by dopaminergic medication and therefore receive STN-DBS as a routine standard of care with routinely collected data.

In total 110 patients who are candidates for STN-DBS will be enrolled in four participating sites in Switzerland and the EU.

ELIGIBILITY:
Inclusion Criteria:

For all subjects:

* Informed consent as documented by signature
* Diagnosis of PD based on the MDS clinical diagnostic criteria for Parkinson's disease
* Fulfilling criteria for STN-DBS:
* The presence of disabling motor complications of dopaminergic treatment
* The absence of surgical contraindications
* Planned bilateral STN-DBS using steering electrodes in the next 3 months (routine standard of care)

Exclusion Criteria:

* Presence of dementia as indicated by a score ≤ 25 on the MOntreal Cognitive Assessment (MOCA)
* Depression with acute suicidal ideation
* Presence of major ongoing psychiatric illness
* Non-compensated systemic disease (i.e., diabetes, hypertension)
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Participation in interventional trial within the 30 days preceding and during the present study
* Previous enrolment into the current study
* Enrolment of any study site personnel, their family members, employees or other dependent persons

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The project population consists of PD patients suffering from levodopa-responsive PD which are not adequately controlled by dopaminergic medication and therefore receive STN-DBS as a routine standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of non-motor fluctuations | Follow-up ≤ 5 Weeks
  Evaluation of the Neuropsychiatric Fluctuations Scale (NFS) in different states (ON/OFF) to evaluate if non-motor fluctuations are present. The bigger the difference between the two subscores ('ON psychological state' and 'OFF psychological sate') in the different states are, the more non-motor fluctuations are present.

SECONDARY OUTCOMES:
Evaluation of motor improvement | Follow-up ≤ 5 Weeks
  Motor improvement following STN-DBS using the Vercise directional leads will be assessed by comparing MDS-UPDRS III score (International Parkinson and Movement Disorder Society) during the study in different states (ON/OFF). The minimum and maximum values are: 0-132, where a higher score means a worse outcome.
Evaluation of STN-DBS induced dysarthria | Follow-up ≤ 5 Weeks
  Dysarthria will be measured during the study by Voice Handicap Index 30 (VHI) scale. The minimum and maximum values are: 0-120, where a higher score means a worse outcome.
Evaluation of postoperative apathy | Follow-up ≤ 5 Weeks
  Apathy will be measured during the study by Dimensional Apathy Scale (DAS). The minimum and maximum values are: 0-72, where a higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ines Debove, MD, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (4):
- France (2):
  - Hospices Civils de Lyon (Centre Hospitalier Universitaire de Lyon), Lyon
  - Hôpital Pitié-Salpêtrière, Paris
- Universitätsklinikum Würzburg, Würzburg, Germany
- Insel Gruppe AG University Hospital Bern, Bern, Switzerland